CLINICAL TRIAL: NCT01764594
Title: A Multicenter, Investigator- and Subject-Blind, Randomized, Placebo-Controlled, Parallel-Group, Repeat-Dose Study to Evaluate the Effect of CDP7657 in Subjects With Active Systemic Lupus Erythematosus
Brief Title: Safety Study of CDP7657 in Patients With Systemic Lupus Erythematosus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Collaborators: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: SL0014; 2012-000631-11 (EudraCT Number)
Record Dates: First submitted 2013-01-02; First posted 2013-01-09 (Estimated); Last update posted 2015-07-16 (Estimated); Status verified 2015-07

CONDITIONS: Immune System Diseases; Autoimmune Diseases; Lupus Erythematosus, Systemic; Skin and Connective Tissue Diseases; Connective Tissue Disease
Keywords: Lupus; SLE
MeSH Terms: conditions — Immune System Diseases; Autoimmune Diseases; Lupus Erythematosus, Systemic; Skin and Connective Tissue Diseases; Connective Tissue Diseases | interventions — dapirolizumab pegol

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CDP7657 (Experimental): CDP7657 100 mg/ ml solution
  30 mg/ kg initial dose
  15 mg/ kg every other week
  10 weeks
  Interventions: Biological: CDP7657
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: CDP7657 — CDP7657 100 mg/ ml solution
  30 mg/ kg initial dose
  15 mg/ kg every other week
  10 weeks
  Arms: CDP7657
Other: Placebo — Placebo comparator
  Arms: Placebo

SUMMARY:
To evaluate safety, tolerability pharmacokinetics and immunogenicity of CDP7657.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Systemic Lupus Erythematosus (SLE)

Exclusion Criteria:

* Severe neuropsychiatric or severe renal Systemic Lupus Erythematosus (SLE)
* History of chronic, recurrent, or recent severe infection
* Significant hematologic abnormalities
* History of cancer, heart failure, renal disease, liver disease or other serious illness

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-01; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with at least one Treatment-emergent Adverse Event (TEAE) during the study | 0 - 28 Weeks
Percentage of subjects who withdrew due to an Treatment-emergent Adverse Event (TEAE) during the study | 0 - 28 Weeks

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) | 0 - 28 Weeks
Predose plasma concentration (Ctrough) | 0 - 28 Weeks
Area under the concentration-time curve over the dosing interval (AUCτ) | 0 - 28 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493
Locations (21):
- Belgium (2):
  - 102, Brussels
  - 101, Leuven
- Bulgaria (3):
  - 203, Plovidv
  - 201, Sofia
  - 202, Sofia
- Germany (6):
  - 301, Berlin
  - 303, Erlangen
  - 305, Frankfurt
  - 306, Greifswald
  - 304, Hanover
  - 302, Kiel
- Poland (2):
  - 501, Krakow
  - 503, Wroclaw
- Romania (2):
  - 601, Bucharest
  - 602, Cluj-Napoca
- Russia (2):
  - 701, Moscow
  - 702, Yaroslavl
- Spain (4):
  - 401, Hospitalet Del Llobregat
  - 402, Santiago de Compostela
  - 404, Seville
  - 405, Seville

REFERENCES:
- [Derived] Chamberlain C, Colman PJ, Ranger AM, Burkly LC, Johnston GI, Otoul C, Stach C, Zamacona M, Dorner T, Urowitz M, Hiepe F. Repeated administration of dapirolizumab pegol in a randomised phase I study is well tolerated and accompanied by improvements in several composite measures of systemic lupus erythematosus disease activity and changes in whole blood transcriptomic profiles. Ann Rheum Dis. 2017 Nov;76(11):1837-1844. doi: 10.1136/annrheumdis-2017-211388. Epub 2017 Aug 5. PMID 28780512